CLINICAL TRIAL: NCT03564990
Title: The Impact of Interactive, Multifaceted Approach Education on Parental Anxiety, Knowledge and Satisfaction for Congenital Cataract: A Randomized, Controlled Trial
Brief Title: The Impact of Interactive, Multifaceted Approach Education on Congenital Cataract
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Haotian Lin, Prof., Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CCPMOH2018-China-3
Record Dates: First submitted 2018-06-05; First posted 2018-06-21 (Actual); Last update posted 2018-06-21 (Actual); Status verified 2018-06

CONDITIONS: Congenital Cataract
MeSH Terms: interventions — Drug Interactions

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- interactive, multifaceted approach (Experimental): A health education module consisting of a lecture and workshop was incorporated into a health-care course.
  Interventions: Other: interactive, multifaceted approach
- conventional approach (Sham Comparator): conventional follow-up with oral healthy education
  Interventions: Other: conventional approach

INTERVENTIONS:
Other: interactive, multifaceted approach — A health education module consisting of a lecture and workshop was incorporated into a health-care course.
  Arms: interactive, multifaceted approach
Other: conventional approach — conventional follow-up
  Arms: conventional approach

SUMMARY:
To evaluate the impact of a health education program on parental anxiety, the comprehension-memorization of the information and their satisfaction.

DETAILED DESCRIPTION:
Prospective study including parents of congenital cataract, randomized in two groups: health education program with an interactive, multifaceted approach versus conventional follow-up. A health education module consisting of a lecture and workshop was incorporated into a health-care course. A non-validated survey assessed knowledge. Parental stress was assessed using self-questionnaires before and after training .At each moment we evaluated the level of anxiety, satisfaction of information quality and the comprehension-memorization of the data.

ELIGIBILITY:
Inclusion Criteria:

* children with regulated cataract surgery

Exclusion Criteria:

* difficulty in understanding the language
* uncompleted questionnaires or badly filled in by two different people

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-06-30 (Estimated); Primary Completion 2018-07-30 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
Parenting stress | 12 months
  Parenting stress was assessed using the Parenting Stress Index (PSI)

CONTACTS AND LOCATIONS:
Overall Officials: Haotian Lin, Ph.D, Principal Investigator — Professor
Locations (1):
- Zhognshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China